CLINICAL TRIAL: NCT03998215
Title: Immunogenicity of Diphtheria Booster Vaccination in Adolescents With Inflammatory Bowel Disease
Brief Title: Diphtheria Vaccination in Adolescents With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Wroclaw Medical University (Other); Poznan University of Medical Sciences (Other); Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Lukasz Dembinski, Principal Investigator, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dembinski2012
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Diphtheria; Inflammatory Bowel Diseases
MeSH Terms: conditions — Diphtheria; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diphtheria booster vaccination (Experimental): One booster dose of the trivalent vaccine against diphtheria, tetanus and acellular pertussis
  Interventions: Biological: Diphtheria booster vaccination

INTERVENTIONS:
Biological: Diphtheria booster vaccination — Participants received intramuscularly in the deltoid muscle one dose of the trivalent vaccine against diphtheria, tetanus and acellular pertussis

SUMMARY:
Assessment of the immunogenicity and safety of booster immunization against diphtheria in children with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn's disease or ulcerative colitis based on standard clinical, endoscopic, histologic and radiographic criteria (Porto criteria),
* vaccination, as a part of the basic vaccination course, with five doses of diphtheria, tetanus and whole-cell pertussis vaccine, without booster dose after the age of 6,
* written consent of the patient's legal guardians and the patient himself if he/she turns 16 years of age.

Exclusion Criteria:

* serious exacerbation of inflammatory bowel disease defined as Paediatric Ulcerative Colitis Activity Index (PUCAI) > 65 points for patients with ulcerative colitis or Pediatric Crohn's Disease Activity Index (PCDAI) > 40 points for patients with Crohn's disease.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
Achieving seroprotective antibody concentration | after 4-8 weeks
  Antibody concentrations ≥0.1 IU/ml indicated protection against diphtheria, while levels ≥1.0 IU/ml were considered to ensure long-term protection.

SECONDARY OUTCOMES:
Booster response | after 4-8 weeks
  Booster response was defined as a post-vaccination antibody concentration ≥0.4 IU/mL in initially seronegative subjects or as a fourfold increase of antibody concentration in initially seropositive ones.
Adverse effects | 3 days
  Evaluation of adverse effects after vaccination.
Inflammatory bowel disease exacerbation occurrence. | after 4-8 weeks
  Disease exacerbation assessed according to the Paediatric Ulcerative Colitis Activity Index (PUCAI) for patients with ulcerative colitis or Pediatric Crohn's Disease Activity Index (PCDAI) for patients with Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Banaszkiewicz, MD, PhD, Study Director — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dembinski L, Krzesiek E, Klincewicz B, Grzybowska-Chlebowczyk U, Demkow U, Banaszkiewicz A, Radzikowski A. Immunogenicity of Diphtheria Booster Vaccination in Adolescents With Inflammatory Bowel Disease. Pediatr Infect Dis J. 2020 Mar;39(3):244-246. doi: 10.1097/INF.0000000000002547. PMID 32032309